CLINICAL TRIAL: NCT01406678
Title: Effect of Remote Ischemic Preconditioning in Patients Undergoing On-pump Coronary Artery Bypass Graft Surgery With Crystalloid Cardioplegic Arrest
Brief Title: Remote Ischemic Preconditioning in Coronary Artery Bypass Grafting With Cold Crystalloid Cardioplegic Arrest
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Matthias Thielmann, Matthias Thielman, MD, PhD, University Hospital, Essen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WDHZ-TC-0801
Record Dates: First submitted 2009-12-01; First posted 2011-08-01 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Myocardial Injury
Keywords: remote ischemic preconditioning; coronary artery bypass grafting; myocardial injury
MeSH Terms: interventions — Coronary Artery Bypass; Isoflurane; Sufentanil

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RIPC (Active Comparator): Remote ischemic preconditioning (RIPC) protocol before coronary artery bypass surgery consists of 3 cycles of 5 minutes left upper arm ischemia by inflation of a blood pressure cuff to 200 mmHg and 5 minutes of reperfusion after induction of anesthesia before coronary artery bypass surgery. For myocardial molecular analyses, left ventricular biopsies are taken before induction of cardioplegic cardiac arrest and 5 and 10 Minutes after aortic unclamping during reperfusion of the myocardium.
  Interventions: Procedure: RIPC; Drug: isoflurane+sufentanil anesthesia
- Control (Placebo Comparator): Control group: Coronary artery bypass surgery without remote ischemic preconditioning protocol
  Interventions: Procedure: Control; Drug: isoflurane+sufentanil anesthesia

INTERVENTIONS:
Procedure: RIPC — 3 cycles of 5 min left upper arm ischemia by inflation of a blood pressure cuff to 200 mmHg and 5 min reperfusion
  Other Names: RIPC: Remote ischemic preconditioning; CABG: Coronary artery bypass grafting
  Arms: RIPC
Procedure: Control — Coronary artery bypass surgery without remote ischemic preconditioning protocol
  Other Names: Coronary artery bypass surgery
  Arms: Control
Drug: isoflurane+sufentanil anesthesia — Anaesthesia is maintained by inhaled isoflurane in concentrations 0.7-0.8 % end-tidal with additional sufentanil injected during surgery, as required. During extracorporal circulation patients receive isoflurane via a vaporizer incorporated in the extracorporeal gas supply in the same concentrations.
  Other Names: Isoflurane, (2-chloro-2-(difluoromethoxy)-1,1,1-trifluoro-ethane), Forane; Sufentanil, Sufenta, (R-30730)

SUMMARY:
Remote ischemic preconditioning (RIPC) with transient upper limb ischemia/reperfusion reduces myocardial injury in patients undergoing on-pump coronary artery bypass (CABG) surgery with cross-clamp fibrillation or blood cardioplegia for myocardial protection. The present study assesses protection of heart, brain and kidney by RIPC under crystalloid cardioplegic arrest. The study also addresses safety and clinical outcome.

DETAILED DESCRIPTION:
Remote ischemic preconditioning (RIPC) protocol after induction of anesthesia and before skin incision consists of 3 cycles of 5 minutes left upper arm ischemia by inflation of a blood pressure cuff to 200 mmHg and 5 minutes of reperfusion. For myocardial molecular analyses, left ventricular biopsies are taken before induction of cardioplegic cardiac arrest and at 10 minutes after aortic unclamping during reperfusion of the myocardium.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients >18 years of age
* Double- or triple-vessel coronary artery disease
* Elective isolated first-time CABG
* Combined valve surgery + CABG
* Written informed consent

Exclusion Criteria:

* Renal failure (creatinine ≥ 200 µmol/L)
* Peripheral vascular disease affecting upper limbs
* Preoperative inotropic support
* Any kind of mechanical assist device
* Acute or recent (<4 weeks) acute coronary syndromes
* Any PCI (<6 weeks)
* Any reasons for preoperative cTnI elevation
* Emergency surgery
* Redo surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1204 (Actual)
Dates: Start 2008-07; Primary Completion 2018-03 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Perioperative extent of myocardial injury as measured by cardiac troponin I serum release over 72 hours after CABG surgery and its area under the curve (AUC). | 72 hours postoperatively after CABG surgery

SECONDARY OUTCOMES:
All-cause mortality | 30 days and 1 year and complete follow-up after CABG surgery
Major adverse cardiac and cerebrovascular events (MACCE) | at 30 days and 1 year and complete follow-up after CABG surgery
Myocardial infarction | 30 days and 1 year and complete follow-up after CABG surgery
Renal function | 72 hours post CABG

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Thielmann, MD, PhD, Principal Investigator — Department of Thoracic and Cardiovascular Surgery, West-German Heart Center, University Duisburg-Essen, Essen, Germany; Eva Kottenberg, M.D., PhD., Principal Investigator — Klinik für Anästhesiologie und Intensivmedizin, Universität Duisburg-Essen, Universitätsklinikum Essen, Essen, Germany; Gerd Heusch, M.D., PhD., Principal Investigator — Institut für Pathophysiologie, Universität Duisburg-Essen, Universitätsklinikum Essen, Essen, Germany
Locations (1):
- Department of Thoracic and Cardiovascular Surgery, West-German Heart Center, University Duisburg-Essen, Essen, Germany

REFERENCES:
- [Result] Thielmann M, Kottenberg E, Boengler K, Raffelsieper C, Neuhaeuser M, Peters J, Jakob H, Heusch G. Remote ischemic preconditioning reduces myocardial injury after coronary artery bypass surgery with crystalloid cardioplegic arrest. Basic Res Cardiol. 2010 Sep;105(5):657-64. doi: 10.1007/s00395-010-0104-5. Epub 2010 May 21. PMID 20495811
- [Derived] Zhang L, Zhou K, Gu T, Xu J, Shi M, Zhu J, Liu J. Cardiopulmonary Protection of Modified Remote Ischemic Preconditioning in Mitral Valve Replacement Surgery: A Randomized Controlled Trial. Cardiovasc Ther. 2024 Jun 24;2024:9889995. doi: 10.1155/2024/9889995. eCollection 2024. PMID 39742012
- [Derived] Frey UH, Klaassen M, Ochsenfarth C, Murke F, Thielmann M, Kottenberg E, Kleinbongard P, Klenke S, Engler A, Heusch G, Giebel B, Peters J. Remote ischaemic preconditioning increases serum extracellular vesicle concentrations with altered micro-RNA signature in CABG patients. Acta Anaesthesiol Scand. 2019 Apr;63(4):483-492. doi: 10.1111/aas.13296. Epub 2018 Dec 11. PMID 30548252
- [Derived] Kottenberg E, Thielmann M, Kleinbongard P, Frey UH, Heine T, Jakob H, Heusch G, Peters J. Myocardial protection by remote ischaemic pre-conditioning is abolished in sulphonylurea-treated diabetics undergoing coronary revascularisation. Acta Anaesthesiol Scand. 2014 Apr;58(4):453-62. doi: 10.1111/aas.12278. Epub 2014 Feb 18. PMID 24548338
- [Derived] Thielmann M, Kottenberg E, Kleinbongard P, Wendt D, Gedik N, Pasa S, Price V, Tsagakis K, Neuhauser M, Peters J, Jakob H, Heusch G. Cardioprotective and prognostic effects of remote ischaemic preconditioning in patients undergoing coronary artery bypass surgery: a single-centre randomised, double-blind, controlled trial. Lancet. 2013 Aug 17;382(9892):597-604. doi: 10.1016/S0140-6736(13)61450-6. PMID 23953384
- [Derived] Kottenberg E, Musiolik J, Thielmann M, Jakob H, Peters J, Heusch G. Interference of propofol with signal transducer and activator of transcription 5 activation and cardioprotection by remote ischemic preconditioning during coronary artery bypass grafting. J Thorac Cardiovasc Surg. 2014 Jan;147(1):376-82. doi: 10.1016/j.jtcvs.2013.01.005. Epub 2013 Mar 1. PMID 23465551
- [Derived] Kleinbongard P, Thielmann M, Jakob H, Peters J, Heusch G, Kottenberg E. Nitroglycerin does not interfere with protection by remote ischemic preconditioning in patients with surgical coronary revascularization under isoflurane anesthesia. Cardiovasc Drugs Ther. 2013 Aug;27(4):359-61. doi: 10.1007/s10557-013-6451-3. No abstract available. PMID 23440355
- [Derived] Heusch G, Musiolik J, Kottenberg E, Peters J, Jakob H, Thielmann M. STAT5 activation and cardioprotection by remote ischemic preconditioning in humans: short communication. Circ Res. 2012 Jan 6;110(1):111-5. doi: 10.1161/CIRCRESAHA.111.259556. Epub 2011 Nov 23. PMID 22116817
- [Derived] Kottenberg E, Thielmann M, Bergmann L, Heine T, Jakob H, Heusch G, Peters J. Protection by remote ischemic preconditioning during coronary artery bypass graft surgery with isoflurane but not propofol - a clinical trial. Acta Anaesthesiol Scand. 2012 Jan;56(1):30-8. doi: 10.1111/j.1399-6576.2011.02585.x. Epub 2011 Nov 21. PMID 22103808